CLINICAL TRIAL: NCT06689332
Title: Improving Quality of Life in Frail, Older Patients with Hematological Cancer Through Geriatric Assessment and Treatment - a Pilot Study
Acronym: IMPROVE pilot
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Odense University Hospital (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: HFE-X 22.18
Record Dates: First submitted 2024-11-12; First posted 2024-11-14 (Actual); Last update posted 2024-11-14 (Actual); Status verified 2024-11

CONDITIONS: Hematological Cancers; Frailty; ELDERLY PEOPLE
Keywords: Pilot study, feasibility study, frailty in hematological cancer, comprehensive geriatric assessment, intervention
MeSH Terms: conditions — Frailty | interventions — Geriatric Assessment

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- Single arm pilot study. Intervention: Comprehensive geriatric assessment. (Experimental): Comprehensive geriatric assessment (CGA) is performed by a geriatrician and a geriatric nurse. CGA in this study includes: Assessment of coexisting diseases and treatments. Review of medications and adjustments as needed. Assessment of symptoms and health related issues including screening for depression, dementia, delirium, nutritional problems, falls, polypharmacy and fatigue. Objective examination including blood tests and electrocardiogram. Assessment of activities of daily living and instrumental activities of daily living through standardized questionnaires. Assessment of domestic conditions, including need for assistance from community-based health care services. Assessment of physical function through history and physical tests. Based on the CGA findings, the geriatrician will initiate relevant interventions (including investigations or treatments) and follow-up as required.
  Interventions: Other: Comprehensive Geriatric Assessment

INTERVENTIONS:
Other: Comprehensive Geriatric Assessment — Comprehensive geriatric assessment (CGA) is performed by a geriatrician and a geriatric nurse. CGA in this study includes: Assessment of coexisting diseases and treatments. Review of medications and adjustments as needed. Assessment of symptoms and health related issues including screening for depression, dementia, delirium, nutritional problems, falls, polypharmacy and fatigue. Objective examination including blood tests and electrocardiogram. Assessment of activities of daily living and instrumental activities of daily living through standardized questionnaires. Assessment of domestic conditions, including need for assistance from community-based health care services. Assessment of physical function through history and physical tests. Based on the CGA findings, the geriatrician will initiate relevant interventions (including investigations or treatments) and follow-up as required.

SUMMARY:
Purpose of the Study This study aims to assess the feasibility of conducting outpatient geriatric health assessment (comprehensive geriatric assessment - CGA) alongside initiation of hematological cancer treatment in frail older adults aged 70 or older, diagnosed with hematological cancer.

Methods This is a pilot study, conducted in preparation for a larger randomized trial (not detailed here). The study will enroll 15 frail patients aged 70 or older, diagnosed with treatment-requiring hematological cancer. Frailty will be assessed using the Geriatric 8 (G8) scoring system, consisting of eight questions, with a score of 14 or below categorizing a patient as frail. Each of the 15 included patients will undergo a CGA concurrently with the start of cancer treatment. This assessment will be conducted by a specialist in geriatric medicine and will include reviews of existing symptoms and comorbidities, cognitive and physical functioning, depressive symptoms, nutritional needs, daily living assistance requirements, and medication usage. The health assessment will involve patient interviews, physical exams, basic physical tests, blood tests, and an electrocardiogram (ECG). Depending on the assessment findings, suitable interventions such as medication adjustments, referrals to physical therapy/rehabilitation, nutritional counseling, or evaluation and treatment for other conditions (e.g., dementia, depression) may be initiated. The geriatric health assessment will not alter the cancer treatment plan.

Study Participants Inclusion Criteria

* Patients aged 70 or older
* Treatment-requiring hematological cancer
* Frailty score (G8) of 14 or lower
* Expected survival > 3 months
* Must be able to understand spoken and written information in Danish. Exclusion Criteria
* Geriatric outpatient consultation within the last 6 months
* Ongoing treatment for another type of cancer, except anti-hormone therapy for stable breast or prostate cancer
* Inability to provide informed consent.

Side Effects, Risks, and Disadvantages The study entails minimal risks and inconveniences. Participants will receive standard hematological cancer treatment and a CGA, a well-established standard procedure within geriatric medicine. A disadvantage may be the need for an additional hospital visit for the CGA. Where feasible, appointments will be coordinated between the hematological and geriatric departments. Additional blood tests and an ECG may also be required if these are not part of the cancer treatment regimen. Minor muscle soreness could occur in participants referred to physical therapy.

Scientific and Ethical Considerations This study is expected to pose minimal inconvenience for participants (mentioned above). The study has the potential to enhance the cancer treatment course for participants by reducing functional decline, improving quality of life, and minimizing treatment side effects, thereby increasing adherence to cancer therapy. Additionally, the study will contribute valuable knowledge for designing a subsequent randomized trial, investigating how to improve cancer treatment and care for older, frail patients with hematological cancers, while preserving their quality of life and functional abilities.

ELIGIBILITY:
Inclusion Criteria:

* Age ≥70 years
* Diagnosis with acute leukemia, chronic myeloid leukemia, chronic lymphocytic leukemia, myelodysplastic syndrome, lymphoma, multiple myeloma, chronic myelomonocytic leukemia or myelofibrosis
* Scheduled systemic cancer treatment or initiated systemic cancer treatment within 6 weeks
* Life expectancy > 3 months
* Geriatric 8 score of ≤14 at screening

Exclusion Criteria:

* Current systemic treatment for other coexisting cancer. Patients receiving anti-hormone treatment for breast- or prostate cancer are not excluded, if no evidence of disease progression (radiological / biochemical) in past 3 months or if treatment is adjuvant.
* Having consulted a geriatric outpatient clinic past 6 months
* Unable to understand Danish
* Unable to give written informed consent

Min Age: 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Enrollment: 17 (Actual)
Dates: Start 2022-09-21 (Actual); Primary Completion 2023-07-03 (Actual); Study Completion 2023-07-03 (Actual)

PRIMARY OUTCOMES:
Inclusion rate | 12 weeks
  succes defined as three participants/month
Completion of intervention | 12 weeks
  Success: 80% of study participants complete CGA within 6 weeks from inclusion
Participant retention | 12 weeks
  Success: ≥80% of study participants complete study activities and 12 weeks of follow-up among partici-pants still alive

CONTACTS AND LOCATIONS:
Overall Officials: Henrik Frederiksen, Consultant, professor, Study Director — Department of Hematology, Odense University Hospital
Locations (1):
- Odense University Hospital, Odense, Odense C, Denmark

IPD SHARING:
Plan to Share IPD: Undecided